CLINICAL TRIAL: NCT02049775
Title: Utility of Narrow Band Endoscopy in Predicting Short and Long Term Risk of Relapse in Patients With Quiescent Ulcerative Colitis
Brief Title: Utilization of NBi in Assessing Luminal INflammaion in IBD (UNBLIND)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UR13/10708
Record Dates: First submitted 2014-01-20; First posted 2014-01-30 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative

ARMS (1):
- NBI (Experimental)
  Interventions: Procedure: NBI

INTERVENTIONS:
Procedure: NBI

SUMMARY:
Ulcerative colitis (UC) is a chronic inflammatory condition of unknown aetiology, characterized by a diffuse confluent mucosal inflammation of the colon starting from the rectum with a relapsing and remitting course. Conventional endoscopy was thought to be a reliable parameter of disease activity, but microscopic inflammation can persist despite normal mucosal findings. Histologically detectable inflammation is associated with a greater risk of subsequent relapse. A flare in UC activity is difficult to predict, but a simple, easily measured biological marker of relapse would be important in guiding the most appropriate therapy.

Recent technological advances in fiber optics, light sources, detectors, and molecular biology have stimulated development of numerous optical methods that promise to significantly improve our ability to evaluate human epithelium in vivo. These methods, collectively termed "optical biopsy," are nondestructive in situ assays of mucosal histopathology using light that can provide instantaneous tissue assessment. Narrow band imaging (NBI) is a novel technique that enhances the diagnostic capability of endoscopes in characterising tissues by using filters in a redgreenblue (RGB) sequential illumination system. This results in improved mucosal contrast and detail.

UC always involves the distal colon and activity is usually greatest in rectosigmoid area. This makes evaluation of the rectum and sigmoid an attractive marker in patients with UC. Unlike serum and faecal markers, endoscopic assessment of the mucosa is unlikely to be affected by systemic disease and would be acceptable test for patients and physicians.

We plan to evaluate THE rectosigmoid mucosa in patients with UC by flexible endoscope using both white light and NBI endoscopy. These patients will be followed by for one year or until they relapse, whichever comes first. The aim of our study is to develop endoscopic biomarkers to predict relapse in acute and quiescent UC.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients referred for lower gastrointestinal endoscopy procedure will be recruited.
* Any age (1885 years), gender or ethnic background
* Able and willing to give an informed consent

Exclusion Criteria:

* Patients known to be intolerant to endoscopy.
* Patients with severe lifethreatening comorbidity as judged by the investigator.
* Patients on therapy with anticoagulation that may preclude taking any biopsies
* Pregnant women or breast feeding mothers
* Patient with toxic megacolon
* patients on medications known to cause bowel inflammation.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2013-04; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Narrow band imaging (NBI) | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospital NHS Trust, Leeds, United Kingdom